CLINICAL TRIAL: NCT00813410
Title: A Single Center, Open-Labeled Exploratory Study to Evaluate a Novel Method for Integrating Insulin Delivery and Glucose Sensing in Subcutaneous Tissue of Type-1 Diabetic Patients
Brief Title: Evaluation of a Novel Method for Integrating Insulin Delivery and Glucose Sensing in Adipose Tissue of Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Univ. Prof. Dr. Thomas Pieber, Medical University Graz, Internal Medicine, Endocrinology and Nuclear Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ZIG96
Record Dates: First submitted 2008-12-20; First posted 2008-12-23 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Glucose measurement at the sc. insulin delivery site — Overnight fasting and oral glucose tolerance test (OGTT) combined with simultaneous subcutaneous insulin delivery and glucose sampling using a single microdialysis or microperfusion probe.

SUMMARY:
The study seeks to use microdialysis and microperfusion techniques to assess the feasibility of performing insulin delivery and glucose sensing at a single subcutaneous tissue site.

DETAILED DESCRIPTION:
Glucose management in type 1 diabetic patients comprises the measurement of glucose in capillary blood obtained by fingersticking and administration of exogenous insulin in the form of a subcutaneous bolus injection or continuous subcutaneous infusion.

The present study seeks to test an alternative treatment approach that combines glucose measurement and insulin delivery at a single subcutaneous tissue site, thereby circumventing the need for fingerstick blood glucose monitoring. Microperfusion and microdialysis probes are applied in type 1 diabetic subjects to perform insulin delivery and glucose sampling at the same adipose tissue site. The feasibility of estimating blood glucose concentrations from the glucose levels measured at the subcutaneous insulin delivery site is then assessed during an overnight fast and an oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus patients aged 18 - 65
* C-peptide negative (≤ 0.05 nmol/L)
* HbA1c (glycosylated haemoglobin A1c) < 10%
* Body Mass Index: 21 - 30 kg/m2
* Informed consent obtained before any trial-related activities.

Exclusion Criteria:

* Severe diabetic complications (e.g., proliferative retinopathy, severe nephropathy)
* Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using adequate contraceptive methods
* Any condition that would interfere with trial participation or evaluation of results, as judged by the investigator
* Treatment with drugs that could interfere with glucose metabolism and subcutaneous insulin absorption
* Subject with mental incapacity or language barriers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
glucose concentration at the subcutaneous insulin delivery site | 20 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD, Principal Investigator — Medical University Graz, Internal Medicine, Endocrinology and Nuclear Medicine
Locations (1):
- Medical University of Graz, Graz, Styria, Austria